CLINICAL TRIAL: NCT05428384
Title: Validation of CardioMEMS HF System Cardiac Output Algorithm IDE
Acronym: VICTOR
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10448
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure; Cardiac Output
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Enrolled Participants: Each participant will have paired CardioMEMS and cardiac MRI measurements at both baseline and 3-month follow-up visits.
  Interventions: Device: MRI/ CardioMEMS comparison

INTERVENTIONS:
Device: MRI/ CardioMEMS comparison — Each subject will have CardioMEMS readings paired with MRI scans

SUMMARY:
The investigation will enroll subjects who have been previously implanted with the CardioMEMS™ Pulmonary Artery Sensor. This clinical investigation is twofold; in the first phase (development phase) data collected will be used to complete development of an algorithm that can estimate cardiac output from CardioMEMS™ Heart Failure (HF) System readings. The second phase (validation phase) of this clinical investigation is intended to compare the Cardiac Output estimate from CardioMEMS HF System to Cardiac Output estimates from Cardiac Magnetic Resonance Imaging (reference standard).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing and able to provide written informed consent prior to any clinical investigation-related procedure.
2. Subject is implanted with the CardioMEMS Pulmonary Artery Sensor for a minimum of 3 months at time of consent.
3. Subject is ≥ 18 years of age.
4. Subject is willing and able to undergo several cardiac Magnetic Resonance Imaging scans. This is including but not limited to:

   * Subject must have all Magnetic Resonance Imaging compatible devices
   * Subject must be able to hold their breath during imaging
   * Subject must be free of all metal bodies, fragments, or implants that would prohibit Magnetic Resonance imaging
5. Subject is willing and able to upload Pulmonary Artery pressure information (i.e., take daily CardioMEMS readings and have their hemodynamic information collected at study visits) and comply with the follow-up requirements.

Exclusion Criteria:

1. Subject will receive or is likely to receive an advanced therapy (e.g., mechanical circulatory support or cardiac transplant) in the next 6 months.
2. Subject was implanted with Cardiac Resynchronization Therapy (CRT)-Pacemaker (CRT-P) or CRT-Defibrillator (CRT-D) for less than 90 days prior to consent.
3. Subject is pregnant or planning to become pregnant in the next 6 months.
4. Subject is enrolled into another trial with an active treatment arm.
5. Subject has significant congenital heart disease that has not been repaired.
6. Subject is implanted with mechanical right heart valve(s).
7. Subject has unrepaired severe valvular disease.
8. Subject has an anticipated life expectancy of < 6 months.
9. Subject has an active, ongoing infection, defined as being febrile, an elevated white blood cell count, on intravenous antibiotics, and/or positive cultures (blood, sputum, or urine).
10. Subject has had a major cardiovascular event (e.g., unstable angina, myocardial infarction, percutaneous coronary intervention, open heart surgery, or stroke, etc.) within 90 days prior to consent.
11. Subject has any condition that, in the opinion of the Investigator, would not allow for utilization of the CardioMEMS HF System to manage the subject using information gained from hemodynamic measurements to adjust medications, including the presence of unexpectedly severe pulmonary hypertension (e.g., trans-pulmonary gradient >15) at implant Right Heart Catheterization, a history of non-compliance, or any condition that would preclude ability to obtain CardioMEMS Pulmonary Artery Sensor readings and paired cardiac Magnetic Resonance Imaging data from being collected.
12. Subjects who, in the opinion of the investigator, are at-risk for serious adverse reaction to Dobutamine (ex. subjects with idiopathic hypertrophic subaortic stenosis and subjects who have shown previous manifestations of hypersensitivity to Dobutamine) should be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This clinical investigation will enroll subjects of all genders who are ≥ 18 years of age from the CardioMEMS HF System patient population. The patient population for this clinical trial consists of potential subjects who have had a CardioMEMS PA Sensor previously implanted for a minimum of 3 months at time of consent.
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Cardiac output estimation | 18 months
  The primary outcome of this clinical investigation is to estimate Cardiac Output from CardioMEMS HF System data. The estimated Cardiac Output will be evaluated for agreement between the CardioMEMS HF System-derived Cardiac Output and the Cardiac Output values from cardiac Magnetic Resonance Imaging in patients with the CardioMEMS HF System

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Piedmont Augusta Hospital, Augusta, Georgia
  - Kansas University Medical Center, Kansas City, Kansas
  - Ascension Providence Hospital, Southfield, Michigan
  - University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
  - St. Francis Hospital, New York, New York
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - Austin Heart, Austin, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT05428384/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT05428384/SAP_001.pdf